CLINICAL TRIAL: NCT04990037
Title: A Phase 1b Dose Escalation and Expansion Study of CAN04, a Monoclonal Antibody Targeting IL1RAP, in Combination With Modified FOLFIRINOX in Subjects With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: A Study of the Safety and Tolerance of CAN04 in Combination With FOLFIRINOX in Subjects With Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: CAPAFOUR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cantargia AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN04CLIN003
Record Dates: First submitted 2021-06-21; First posted 2021-08-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Carcinoma; Adenocarcinoma; Pancreatic Cancer; Metastatic
MeSH Terms: conditions — Carcinoma; Adenocarcinoma; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAN04 and FOLFIRINOX (Experimental): Subjects will receive bi-weekly doses of CAN04 in combination with FOLFIRINOX given as standard regimen.
  Interventions: Drug: CAN04; Drug: FOLFIRINOX

INTERVENTIONS:
Drug: CAN04 — Administered intravenously
  Other Names: Nadunolimab
Drug: FOLFIRINOX — Administered intravenously

SUMMARY:
This study will consider the safety and effectiveness of a study drug, CAN04, in combination with FOLFIRINOX, in the treatment of metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The subject is capable to understand and willing to provide written informed consent before any study-related activities (study-related activities are any procedures that would not have been performed during normal management of the subject's disease).
* The subject is at least 18 years of age.
* The subject has been diagnosed with stage IV PDAC (Pancreatic Ductal Adenocarcinoma) and is amenable to first-line systemic therapy. The subject must have measurable disease that is histologically or cytologically confirmed.
* The subject has an ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
* The subject has a primary or metastatic lesion amenable to biopsy and is willing to undergo repeat biopsies, unless a biopsy would not be safe in the opinion of the investigator and in agreement by the sponsor and medical monitor (or designee).
* The subject has clinically adequate bone marrow, hepatic, and renal function based on clinical laboratory test values at screening within the following ranges:

  * Creatinine clearance >30 mL/min calculated by Cockcroft-Gault formula
  * Haemoglobin >90 g/L (blood transfusions during the screening period are not allowed)
  * Absolute neutrophil count >1.5 × 109/L (usage of growth factors, such as G-CSF (Granulocyte Colony-Stimulating Factor), during the screening period is not allowed)
  * Platelets >100 × 109/L
  * Total bilirubin <1.5 × ULN unless due to Gilbert's syndrome
  * AST and ALT ≤3 × ULN (or <5 × ULN for subjects with hepatic metastases)
* The subject has a QT interval corrected using Fridericia's formula (QTcF) of ≤ 480 milliseconds at screening.
* Female subjects of childbearing potential (more info can be found in the protocol) and male subjects with female partners of childbearing potential must be willing to adhere to contraceptive requirements as detailed in the protocol, from at least 1 month prior to study entry to at least 4 months after the last dose of study treatment.
* The subject has suitable venous access for safe drug administration and the study- required drug concentration and pharmacodynamic sampling.

Exclusion Criteria:

* Subjects who have received previous radical radiotherapy, chemotherapy, or investigational therapy for the treatment of metastatic disease.

  * Prior treatment with 5-FU or gemcitabine administered as a radiation sensitiser during and up to 4 weeks after radiation therapy, is allowed; however, if there is lingering toxicity (Grade >1), then the sponsor should be consulted.
  * If a subject received adjuvant or neoadjuvant chemotherapy, tumour recurrence or disease progression must have occurred no sooner than 6 months after completing the last dose.
* Subjects with uncontrolled brain metastases; however, subjects are allowed if they have been previously treated with surgery, whole-brain radiation, and/or stereotactic radiosurgery and are considered controlled (with ≤10 mg/day of prednisone or equivalent) at the time of receiving the first dose of CAN04. For asymptomatic subjects, screening brain imaging is not required.
* Subjects with endocrine or acinar pancreatic carcinoma.
* Subjects with an active severe infection requiring parenteral antibiotics at the time of enrolment or subjects currently receiving oral antibiotics as a continuation of a previous course of parenteral antibiotics.
* Subjects with peripheral sensory neuropathy Grade ≥2.
* Subjects with a serious uncontrolled medical disorder that, in the opinion of the investigator or medical monitor, makes it unwise for the subject to participate in the study or that might jeopardise compliance with the protocol.
* Subjects with psychiatric illness/social circumstances that would limit compliance with study requirements and substantially increase the risk of AEs (Adverse Events) or has compromised ability to provide written informed consent.
* Subjects with an active second invasive malignancy with the exception of stable prostate cancer on watchful waiting.
* Subjects with uncontrolled or significant cardiovascular disease defined as NYHA (New York Heart Association) classification III or IV.
* Subjects with congenital long QT syndrome.
* Subjects with a history of autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day).
* Subjects with known hepatitis B virus surface antigen seropositive or detectable hepatitis C infection viral load. NOTE: Subjects who have positive hepatitis B core antibody or hepatitis B surface antigen antibody can be included but must have an undetectable hepatitis B viral load.
* Subjects with a known history of any other relevant congenital or acquired immunodeficiency other than HIV infection. NOTE: Subjects testing positive for HIV are NOT excluded from this study, but HIV- positive subjects must meet the following criteria:

  * Have CD4+ T-cell (CD4+) counts ≥350 cells/µL.
  * Have not had an opportunistic infection within the past 12 months. Subjects on prophylactic antimicrobials can be included in the study.
  * Should be on established antiretroviral therapy for at least 4 weeks.
  * Have an HIV viral load less than 400 copies/mL prior to enrolment.
* Subjects who receive a live vaccination, etanercept, or other TNF-α (Tumor Necrosis Factor-alpha) inhibitors during or just prior to (within 28 days of first dose of study treatment) participation in this study.
* Subjects who have had a hospitalization for bowel obstruction within 12 weeks prior to enrolment.
* Subjects with a known bleeding disorder or coagulopathy. NOTE: Subjects on stable anticoagulant therapy are allowed at the discretion of the investigator; however, these subjects should be monitored more frequently.
* Subjects with a known or suspected allergy to any study treatment or related products, including platinum-based chemotherapeutic agents.
* Female subjects who are pregnant or breastfeeding or trying to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Frequency of TEAEs (Treatment-emergent adverse events) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Number of participants with DTLs (dose-limiting toxicities) | Up to day 28
Number of subjects with 1 or more TEAEs leading to dose modifications | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Number of subjects with grade ≥ 3 TEAEs | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Percentage of subjects with grade ≥ 3 TEAEs | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Number of subjects with 1 or more TEAEs leading to treatment discontinuation | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Percentage of subjects with 1 or more TEAEs leading to dose modification | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Percentage of subjects with 1 or more TEAEs leading to treatment discontinuation | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Number of subjects with 1 or more SAEs (serious adverse events) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Percentage of subjects with 1 or more SAEs | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.

SECONDARY OUTCOMES:
Serum Concentrations of CAN04 and Folfirnox | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Antidrug antibodies (ADAs) against CAN04 | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Change in serum IL-6 (Interleukin-6) concentration | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Change in serum CRP (C-reactive protein) concentration | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Overall response rate (ORR) | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
  Proportion of subjects with partial response (PR) or complete response (CR) to study treatment as defined by iRECIST (immune-related response evaluation criteria in solid tumors) and measured by radiological assessment (CT/MRI Scan)
Progression free survival | From the first dose until the last subject has completed their end of trial visit or the last enrolled subject has completed 6 months of treatment, whichever comes first.
Overall Survival | Up to 36 months after 1st dose of last subject (or death)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia-Ribas, MD, PhD, Study Director — Cantargia AB
Locations (9):
- France (4):
  - EDOG - Institut Bergonie - PPDS, Bordeaux
  - EDOG Institut de Cancerologie de l'Ouest - PPDS, Nantes
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
- Spain (5):
  - Instituto de Investigacion Oncologica Vall d'Hebron (VHIO) - EPON, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - START MADRID_Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No